CLINICAL TRIAL: NCT05394935
Title: The Effects of High- and Moderate-Intensity Exercise on the Cerebrovascular and Cardiometabolic Health of Women With Polycystic Ovary Syndrome
Brief Title: The Effects of High-intensity and Moderate-intensity Exercise on Polycystic Ovary Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cardiff Metropolitan University (Other)
Collaborators: Cardiff University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: STA-1653
Record Dates: First submitted 2022-02-10; First posted 2022-05-27 (Actual); Last update posted 2025-02-13 (Actual); Status verified 2025-02

CONDITIONS: Polycystic Ovary Syndrome; Exercise; Cerebrovascular Circulation
Keywords: PCOS; Polycystic Ovary Syndrome; Exercise; High-Intensity Interval Training; Moderate-Intensity Steady State; Cerebrovascular
MeSH Terms: conditions — Polycystic Ovary Syndrome; Motor Activity | interventions — High-Intensity Interval Training

STUDY DESIGN:
Intervention Model Description: Participants will complete multiple baseline assessments. Within the crossover model, participants will complete a baseline cerebrovascular assessment, followed by a random bout of acute exercise and then a post-exercise repeat of the baseline tests. Following a pre-designated washout, the participants will complete the same visit with the remaining exercise bout.
Who Masked: Outcomes Assessor
Masking Description: All participant data and exercise arm will be anonymised and non-identifiable by the assessor.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Polycystic Ovary Syndrome (Experimental): Women with PCOS
  Interventions: Other: High-Intensity Exercise; Other: Moderate-Intensity Exercise
- Controls (Active Comparator): Healthy, age and BMI matched controls
  Interventions: Other: High-Intensity Exercise; Other: Moderate-Intensity Exercise

INTERVENTIONS:
Other: High-Intensity Exercise — Acute, low-volume HIIT 12x (1min:1min) Working intensity: >85% heart rate reserve Resting intensity: Active rest
Other: Moderate-Intensity Exercise — Continuous, MISS 50mins Working intensity: 50-60% heart rate reserve

SUMMARY:
This study will investigate the impact of high- and moderate-intensity exercise on the cardiometabolic and brain health of women with Polycystic Ovary syndrome (PCOS). The aim is to measure and compare normal, healthy women without PCOS, to those with the condition.

All participants will undergo a blood test. The investigators will then assess the participants cardiovascular fitness by means of a maximal exercise test and measure body composition through height, weight, and hip-to-waist ratio.

Participants will undergo an MRI, where the investigators will assess the participants brain structure and how the brain responds to a number of tests. The investigators will also conduct some tests that will assess the participants cognition, such as IQ, memory etc.

The investigators will measure the blood vessels leading to the brain and the blood flow through them to measure how much blood the brain receives when rested, using ultrasound.

The investigators will use a number of tests to look at brain function, measure the responses to these tests, and compare them between the normal, healthy women and those with PCOS. This will show if women with PCOS have a similar brain function when rested and when their brains are tested to those without the condition.

The investigators will use exercise as an intervention, where the aim will be to investigate whether women with PCOS respond similarly to those without the condition to both high-intensity and moderate-intensity exercise. The tests of brain function will be repeated following the exercise, and see if both normal, healthy women and those with PCOS have a similar response to the brain function tests.

All tests and measures will be compared between the PCOS group, and the healthy control group to establish any potential differences or similarities as a result of the condition.

ELIGIBILITY:
Inclusion Criteria:

* Polycystic Ovary Syndrome as diagnosed by any recognised criteria.
* Inactive (less than 40 mins of structured exercise per week).

Exclusion Criteria:

* Pregnant or breastfeeding.
* Congenital adrenal hyperplasia, Cushing's syndrome, thyroid disease, hyperprolactinaemia and androgen secreting tumours.
* Known history of cardiovascular disease.
* Contraindications to MRI (fitted with ferromagnetic devices).

Ages: 16 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Gender Based: Yes — Females with PCOS and healthy females acting as a controls. Eligibility of participants is via biological sex.
Enrollment: 34 (Actual)
Dates: Start 2020-01-01 (Actual); Primary Completion 2024-05-25 (Actual); Study Completion 2024-05-25 (Actual)

PRIMARY OUTCOMES:
Cerebrovascular Reactivity to Carbon Dioxide (CO2) | Baseline
  6% CO2 administered to measure reactivity of the cerebrovasculature as measured by extra-cranial ultrasonography.
Cerebrovascular Reactivity to Carbon Dioxide (CO2) | Less than 1 hour post-exercise
  6% CO2 administered to measure reactivity of the cerebrovasculature as measured by extra-cranial ultrasonography.
Neurovascular coupling (NVC) | Baseline
  NVC will be assessed using a visual task (flashing checkerboard) measured via transcranial Doppler.
Neurovascular coupling (NVC) | Less than 1 hour post-exercise
  NVC will be assessed using a visual task (flashing checkerboard) measured via transcranial Doppler.
Dynamic cerebral autoregulation (dCA) | Baseline
  dCA will be assessed using a squat-stand method to induce forced oscillations in blood pressure and measured using finger plethysmography and transcranial Doppler.
Dynamic cerebral autoregulation (dCA) | Less than 1 hour post-exercise
  dCA will be assessed using a squat-stand method to induce forced oscillations in blood pressure and measured using finger plethysmography and transcranial Doppler.
Cerebral blood velocity in the middle (MCAv) and posterior cerebral arteries (PCAv) during exercise | During high-intensity exercise (24 minutes)
  MCAv and PCAv will be assessed using transcranial Doppler and employed throughout both bouts of acute exercise.
Cerebral blood velocity in the middle (MCAv) and posterior cerebral arteries (PCAv) during exercise | During moderate-intensity exercise (50 minutes)
  MCAv and PCAv will be assessed using transcranial Doppler and employed throughout both bouts of acute exercise.

SECONDARY OUTCOMES:
Cardiorespiratory fitness (CRF) | Baseline
  CRF will be assessed via peak oxygen uptake using a step protocol on a cycle ergometer. to achieve VO2peak.
Cerebral structure | Baseline
  MRI will be employed to assess grey and white matter structure.
Cerebral blood flow | Baseline
  Functional MRI will be employed to assess global and regional cerebral blood flow.
Cerebral metabolic rate of oxygen consumption | Baseline
  Functional MRI will be employed to assess cerebral metabolic rate of oxygen consumption.
Cerebrovascular reactivity | Baseline
  Functional MRI will be employed to assess cerebrovascular reactivity during a breath hold challenge.
Cognitive testing | Baseline
  A comprehensive cognitive battery will be employed to test across multiple cognitive sub-domains (IQ, working memory, episodic memory, attention and executive function).
Blood pressure during exercise | During High-intensity interval exercise (HIIT) (24 minutes) and Moderate-intensity steady state (MISS) (50 minutes) exercise
  Finger plethysmography will be used to non-invasively monitor systolic and diastolic blood pressure throughout both acute bouts of exercise.
Hormone profile | Baseline
  Hormonal profile will be measured through blood sampling, including androstenedione, sex hormone binding globulin and testosterone. From these values, free androgen index (FAI) will be calculated.
Metabolic profile | Baseline
  Metabolic profile will be measured through blood sampling, including fasting glucose and fasting insulin. From these values, the homeostatic model assessment of insulin resistance (HOMA-IR) will be calculated.
Lipid profile | Baseline
  Lipid profile will be measured through blood sampling, including total cholesterol, high-density lipoproteins, low-density lipoproteins and triglycerides.

CONTACTS AND LOCATIONS:
Locations (1):
- Cardiff Metropolitan University, Cardiff, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Applications for access to study- and participant-level data will be considered on direct enquiry.
Supporting Information: Analytic Code
Time Frame: January 2024 - 5 years